CLINICAL TRIAL: NCT00911261
Title: An Open-Label Long Term Effectiveness and Safety Study of Oxymorphone Extended Release Tablets in Patients With Cancer or Neuropathic Pain
Brief Title: Oxymorphone Extended Release in Patients With Cancer or Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, CR&D, Endo Pharmaceuticals Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3202-029
Record Dates: First submitted 2009-05-15; First posted 2009-06-01 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Pain; Neuropathic Pain; Cancer
Keywords: Cancer Pain; Neuropathic Pain; Extended Release; Long-Acting Opioid; Oxymorphone
MeSH Terms: conditions — Chronic Pain; Neuralgia; Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Oxymorphone Extended Release

INTERVENTIONS:
Drug: Oxymorphone Extended Release — * Study Medication: Oxymorphone ER 5 mg, 10 mg, 20 mg, and 40 mg tablets
  * Rescue Medication: Oxymorphone IR 5 mg and 10 mg tablets
  * Treatment will consist of up to 12 months of dosing with Oxymorphone ER.

SUMMARY:
The purpose of this study is to determine if Oxymorphone Extended Release is effective and safe in treating chronic pain in patients with cancer or neuropathic pain.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the analgesic effectiveness and tolerability of oxymorphone ER in the treatment of cancer or neuropathic pain. Opioid-naïve subjects are gradually titrated from oxymorphone ER 5 mg, every 12 hours (q12h). All other subjects are titrated to a stable dose (defined as pain scores ≥ 4 on BPI Question 5 on 3 of 5 consecutive days while receiving the same total daily dose of study medication including rescue) with tolerable side effects. Subjects could potentially receive therapy for up to 12 months after the first dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age or older, with moderate to severe chronic malignant and/or neuropathic pain of at least 3 months duration and either:

  1. have an initial pain intensity score of greater than 4 on a 10-point scale using BPI Question 5, if sub-optimally responding to their current analgesic regimen, or
  2. have intolerable side effects to one or more components of their current opioid-containing analgesic regimen.
* Currently receive a stable (at least 2 weeks duration) analgesic regimen
* If female, must be practicing abstinence or using a medically acceptable form of contraception (e.g., intrauterine device, hormonal birth control, or double barrier method).
* Understand written and spoken English
* Have been informed of the nature of the study and provided written informed consent

Additional Inclusion Criteria for Cancer Patients Only:

* Have a life expectancy of at least 12 months

Additional Inclusion Criteria for Neuropathic Patients Only:

* Have a diagnosis of:

  * post-herpetic neuralgia (PHN)
  * diabetic neuropathy (DN)
  * complex regional pain syndrome (CRPS)
  * HIV neuropathy
  * idiopathic sensory neuropathy
  * traumatic peripheral neuropathy
  * central neuropathic pain condition (spinal cord injury, post-stroke pain), OR
  * other peripheral neuropathy (upon mutual agreement of the sponsor and investigator).

Exclusion Criteria:

* Have a positive pregnancy test (females only)
* Have a history of or active asthma or emphysema
* Have clinically significant hepatic impairment
* Have a history of alcohol or substance abuse within the last 3 years
* Have a history of opioid abuse within 6 months prior to study entry
* Have a known allergy or significant reaction to opioids, including codeine
* Have a known oxymorphone sensitivity or allergy
* Have received an investigational drug or product or participated in an investigational drug study within a period of 30 days prior to receiving study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2003-08; Primary Completion 2005-03 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Tolerability | Throughout the study

SECONDARY OUTCOMES:
Average daily pain intensity (Question 5 of BPI) | Week 1-4, Month 12
Question 3, 4, 5, 6, 8, and 9 of BPI questionnaire | Week 1-4, Month 12
Average daily dose of oxymorphone ER | Daily
Average daily dose of rescue medication | Daily
Total daily dose of oxymorphone ER and rescue medication | Daily
Time to stabilization | Month 12
Patient/investigator global assessment of pain relief | Month 12
Treatment Satisfaction | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals